CLINICAL TRIAL: NCT07262606
Title: Salivary Mitofusin-1 Levels in Periodontitis: Associations With Disease Severity, Smoking, and Treatment Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer Faruk Okumuş (Other)
Responsible Party: Sponsor-Investigator, Ömer Faruk Okumuş, assistant professor, Erzincan University
Organization: Erzincan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EBYU-OKUMUS-MFN1-2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Disease; Chronic Periodontitis (Disorder)
Keywords: Mitofusin-1; Saliva; Biomarker; Periodontal Treatment; Smoking
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis; Smoking | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Control Group (Sham Comparator): Periodontally healthy individuals with no clinical attachment loss, probing depth ≤3 mm, no radiographic bone loss, and low gingival and plaque index scores.
  Interventions: Other: Saliva Collection
- Mild Periodontitis Group (Experimental): Non-smoking individuals diagnosed with Stage I-II periodontitis according to the AAP/EFP 2018 classification, with clinical attachment loss of 1-4 mm and ≤15-33% radiographic bone loss.
  Interventions: Procedure: Non-surgical Periodontal Therapy (Scaling and Root Planing); Other: Saliva Collection
- Severe Periodontitis Group (Experimental): Non-smoking individuals diagnosed with Stage III-IV periodontitis according to the AAP/EFP 2018 classification, with clinical attachment loss ≥5 mm and radiographic bone loss to the mid-advanced level of the root.
  Interventions: Procedure: Non-surgical Periodontal Therapy (Scaling and Root Planing); Other: Saliva Collection
- Severe Periodontitis with Smoking Group (Experimental): Individuals who meet the criteria for the Severe Periodontitis Group and are also regular smokers (at least 10 cigarettes per day for a minimum of 5 years).
  Interventions: Procedure: Non-surgical Periodontal Therapy (Scaling and Root Planing); Other: Saliva Collection

INTERVENTIONS:
Procedure: Non-surgical Periodontal Therapy (Scaling and Root Planing) — A standard periodontal treatment procedure that involves the removal of dental plaque and calculus (tartar) from the tooth surfaces and root pockets. This is followed by root planing to smooth the root surfaces, allowing the gingiva to heal and reattach to the tooth.
  Arms: Mild Periodontitis Group; Severe Periodontitis Group; Severe Periodontitis with Smoking Group
Other: Saliva Collection — Collection of unstimulated whole saliva. Participants will be asked to allow saliva to pool in the floor of the mouth and then passively drool into a sterile collection tube. A total of 1.5 ml of saliva will be collected from each participant.

SUMMARY:
Periodontitis (gum inflammation) is a common disease worldwide. This study aims to investigate a novel biomarker, a protein called Mitofusin-1 (Mfn1), in saliva that may be associated with the severity of periodontitis and response to treatment. The study will include periodontally healthy individuals, individuals with mild to severe periodontitis, and smokers with severe periodontitis. Participants will receive saliva samples and undergo clinical periodontal examinations. Individuals with periodontitis will receive standard periodontal treatment, and changes in Mfn1 levels will be assessed 3 months after treatment. The study is expected to shed light on the potential utility of Mfn1 as a marker in the diagnosis and follow-up of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Systemically healthy (no history of diabetes mellitus, immunodeficiency, malignancy, or other systemic conditions that could affect periodontal status).
* Have a minimum of 20 natural teeth (excluding third molars).
* No antibiotic therapy or periodontal treatment in the last 6 months.

For Healthy Control Group:

No clinical attachment loss. Probing depth ≤ 3 mm. No radiographic evidence of bone loss. Low gingival and plaque index scores.

For Mild Periodontitis Group:

Diagnosed with Stage I or II periodontitis according to the 2018 AAP/EFP classification.

Clinical attachment loss of 1-4 mm. Radiographic bone loss of ≤15-33%. Non-smoker.

For Severe Periodontitis Group:

Diagnosed with Stage III or IV periodontitis according to the 2018 AAP/EFP classification.

Clinical attachment loss ≥ 5 mm. Radiographic bone loss to the mid-advanced level of the root. Non-smoker.

For Severe Periodontitis with Smoking Group:

Meets all criteria for the Severe Periodontitis Group. Regular smoker (at least 10 cigarettes per day for a minimum of 5 years).

Exclusion Criteria:

* Fewer than 20 natural teeth (excluding third molars).
* Presence of any systemic disease (e.g., diabetes mellitus, immunological disorders, cancer).
* Use of antibiotics or receiving periodontal treatment in the last 6 months.
* Pregnancy or lactation.
* For non-periodontitis groups (Healthy Control): Any signs of periodontitis.
* For periodontitis groups (all): History of smoking cessation for at least 5 years (must be either a current regular smoker or a never-smoker, depending on the group definition).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Salivary Mitofusin-1 (Mfn1) Concentration at Baseline | Baseline
  Mfn1 protein concentration in saliva measured using ELISA (ng/mL) at baseline in each study group.

SECONDARY OUTCOMES:
Change in Salivary Mfn1 Concentration After Periodontal Therapy | Baseline and 3 months
  Difference in salivary Mfn1 concentration (ng/mL) measured using ELISA at baseline and 3 months after non-surgical periodontal therapy in the periodontitis groups.
Salivary Glutathione Peroxidase (GPx) Concentration | Baseline
  GPx enzyme activity measured in saliva by spectrophotometric colorimetric assay (U/L).
Salivary 8-Hydroxy-2'-Deoxyguanosine (8-OHdG) Concentration | Baseline
  8-OHdG concentration measured in saliva using ELISA (ng/mL).
Correlation Between Salivary Mfn1 Concentration and Probing Depth (PD) | Baseline
  Correlation coefficient (r) between salivary Mitofusin-1 (Mfn1) concentration measured by ELISA (ng/mL) and probing depth measured with a manual periodontal probe (mm).
Correlation Between Salivary Mfn1 Concentration and Clinical Attachment Level (CAL) | Baseline
  Correlation coefficient (r) between salivary Mitofusin-1 (Mfn1) concentration measured by ELISA (ng/mL) and clinical attachment level measured with a manual periodontal probe (mm).
Correlation Between Salivary Mfn1 Concentration and Plaque Index (PI) | Baseline
  Correlation coefficient (r) between salivary Mitofusin-1 (Mfn1) concentration measured by ELISA (ng/mL) and plaque index assessed using the Silness-Löe Plaque Index (%).
Correlation Between Salivary Mfn1 Concentration and Gingival Index (GI) | Baseline
  Correlation coefficient (r) between salivary Mitofusin-1 (Mfn1) concentration measured by ELISA (ng/mL) and gingival index assessed using the Löe-Silness Gingival Index (score).

CONTACTS AND LOCATIONS:
Overall Officials: Ömer F Okumuş, DDS,PhD, Principal Investigator — Erzincan Binali Yıldırım University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Erzincan Binali Yıldırım University Faculty of Dentistry, Erzincan, Erzincan, Turkey (Türkiye)